CLINICAL TRIAL: NCT06076070
Title: GENomic PROfilation for Therapeutic Purposes in SARComas and Molecular Tumor Board (MTB): Retrospective/Prospective Study in Referral Centers
Acronym: PROGEN_SARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Candiolo Cancer Institute - IRCCS (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Istituto Oncologico Veneto IRCCS (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Istituto Ortopedico Rizzoli (Other); Ospedale Pediatrico Bambin Gesù (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Istituti Tumori Giovanni Paolo II (Network); Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: RS1607/21
Record Dates: First submitted 2023-03-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-06

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter noninterventional, translational study, retrospective/prospective designed in order to assess the aptitude to the use of genomic profiling methods for therapeutic purposes and evaluation by the institutional Molecular Tumor Board (MTB) of sarcoma patients with metastatic/locally advanced disease that is inoperable with no viable therapeutic alternatives or with histotypes known to be resistant to available in-label medical treatments and without already therapeutically validated driver mutations.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoma patients of any age (inclusion of centers pediatric)
* Patients with any histotype of soft tissue sarcomas and bone
* Patients at any stage of the treatment pathway for disease that is localized or metastatic/inoperable
* Availability of follow-up data
* Written informed consent (prospective part/patients in follow-up)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multicenter noninterventional, translational study, retrospective/prospective designed in order to assess the aptitude to the use of genomic profiling methods for therapeutic purposes and evaluation by the institutional Molecular Tumor Board (MTB) of sarcoma patients with metastatic/locally advanced disease that is inoperable with no viable therapeutic alternatives or with histotypes known to be resistant to available in-label medical treatments and without already therapeutically validated driver mutations.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Evaluate interest and feasibility in carrying out genomic profilingfor building two databases data collection | Baseline
  Specific center database:
  Existence or otherwise of an MTB in the participating structure, composition of the MTB, methods of access to off-label drugs used by the centre, management of incidental findings.
  Patient specific database:
  Identification code, demographic data (age, ethnic origin), histological diagnosis, date of onset disease, stage of disease, any molecular tests performed to define the histotype diagnosis, adjuvant therapy, number of antineoplastic treatments carried out for the disease advanced, date of last recurrence of disease, molecular profile identified, date of presentation to MTB, type of molecular analysis required by MTB, presence or absence of therapeutic target e description of the target identified if present, type of treatment undertaken following the analysis genomics, method of access to the drug for the specific patient, starting date of treatment on a basis molecular, response to treatment, progression-free survival, overall survival.
Extended molecular profile | Baseline
  Analysis of the inclusion of tissue in FFPE relating to the neoplasm under examination.
  RNA and DNA extraction from FFPE tissue will be performed using the kits dedicated qiagen. The NGS analysis will be carried out using a panel of 500 genes, described as oncogenic drivers, starting from 20 ng of nucleic acid, using preparation reagents of the libraries and for sequencing the OCA PLUS Thermofisher Scientific kit, following the protocols indicated by the manufacturer.
  The same kit allows the evaluation tumor mutational burden (TMB), microsatellite instability (MSI) and gene defects PROGEN_SARC Version no. 2.0 - 14.06.2022 11/15 of homologous recombination (HRR) including loss of heterozygosity (LOH).

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy